CLINICAL TRIAL: NCT04041973
Title: An Open-label Individually Randomised Controlled Trial to Assess the Efficacy of Artemether-lumefantrine Prophylaxis for Malaria Among Forest Goers in Cambodia
Brief Title: Study to Assess Efficacy of Artemether-lumefantrine Prophylaxis Against Forest Malaria in Cambodia (PAL_Cambodia)
Acronym: PAL_Cambodia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Global Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MAL19001
Record Dates: First submitted 2019-04-23; First posted 2019-08-01 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2022-05

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination; Geritol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT arm (Experimental): Artemether-lumefantrine (AL) x 3 days followed by 1 day per week
  Interventions: Drug: Artemether-lumefantrine
- Multivitamin arm (Active Comparator): Multivitamin x 3 days followed by 1 day per week
  Interventions: Dietary Supplement: Multivitamin

INTERVENTIONS:
Drug: Artemether-lumefantrine — One tablet AL contains 20 mg artemether and 120 mg lumefantrine
  The prophylaxis will start with a 3-day course of twice daily AL. This will be followed by 2 doses 8 hours apart on one day per week for up to 3 28-35 day consecutive follow-up periods and for 4 weeks after leaving the forest.
  Arms: ACT arm
Dietary Supplement: Multivitamin — One tablet contains Vitamin-A : 5000 USP units, Vitamin D: 400 USP Units, Ascorbic acid: 75 mg, Thiamine Mononitrate: 2 mg, Riboflavin: 3 mg, Niacin amide: 20 mg.
  The prophylaxis will start with a 3-day course of twice daily AL. This will be followed by 2 doses 8 hours apart on one day per week for up to 3 28-35 day consecutive follow-up periods and for 4 weeks after leaving the forest.
  Arms: Multivitamin arm

SUMMARY:
In the Greater Mekong Subregion (GMS) adults are at highest risk for malaria. The most relevant disease vectors bite during daytime and outdoors which makes forest work a high-risk activity for malaria. The absence of effective vector control strategies and limited periods of exposure during forest visits suggest that chemoprophylaxis could be an appropriate strategy to protect forest workers against malaria.

The investigators propose the use of Artemether-lumefantrine (AL), a drug whose efficacy remains high in the GMS, unlike, for example DHA/piperaquine [20]. The proposed study will help to assess the efficacy and feasibility of prophylaxis to prevent malaria in forest workers, help to identify the optimal regimen, and predict its efficacy in reducing overall transmission. The proposed study is a critical step for future use of chemoprophylaxis to protect forest workers in the GMS against malaria.

Funder: Wellcome Trust of Great Britain grant number 106698/Z/14/Z and 220211.

DETAILED DESCRIPTION:
Summary of trial design

An open-label randomised trial among forest goers comparing the ACT AL with a multivitamin with no antimalarial activity to evaluate the efficacy of prophylaxis, and to better understand high risk groups and locations of malaria transmission.

Artemether-lumefantrine prophylaxis trial

The study of AL versus a multivitamin will be a two-arm randomised open label comparative study. Laboratory assessments of malaria infection at baseline and days 28, 56, and 84 will be performed blind to treatment allocation and incidence of clinical cases during follow-up will be recorded.

Activities/outcomes

The main activity proposed is an in vivo clinical assessment of prophylaxis to prevent malaria in 4400 participant episodes in 50 villages in Stung Treng and Pursat Provinces, Cambodia. The subjects will be randomized in a one-to-one ratio between the ACT AL and a multivitamin preparation with no antimalarial activity.

The study sites have been chosen based on current information on incidence of malaria, known predominance of malaria among forest goers, presence of an established clinical research programme and feasibility to perform the proposed research activities.

Efficacy of AL ACT will be assessed through follow up visits every 28 days during a course of prophylaxis when temperature, symptom questionnaires, brief physical examinations, and malaria parasite PCR, lumefantrine levels, and, in selected individuals, parasite genetics will be performed. Episodes of confirmed clinical malaria among study participants at any time point between enrolment and follow-up will also be recorded.

All the organisations in this collaboration will work closely with local counterparts including the National Malaria Control Programmes (NMCPs), non-governmental and other relevant organisations. Training is an integral part of this collaborative working relationship, and the building of local research capacity is an essential component of all research plans.

All research-related activities, from study design, planning, implementation through to analysis and writing of reports will be performed jointly with local counterparts. Both on-the-job training and formal training will be provided when needed, in particular for Good Clinical Practice (GCP) skills.

The close interaction between WHO and its regional offices will ensure that new knowledge is disseminated efficiently and effectively throughout the region.

Study duration

The recruitment phase of the study is expected to last 12 months following the intended start of recruitment in July 2019. Training and community sensitization will precede study execution for 3 months. Data management and analysis, sample analysis (PCR, parasite genetics, lumefantrine levels), mathematical modelling and report writing are expected to take about 5 months. Therefore, the total time to complete the study will be about 20 months.

ELIGIBILITY:
Inclusion criteria

* Male or female, adults aged between 16 and 65 years.
* Planning to travel to the forest within the next 72 hours and stay overnight.
* Written informed consent.
* Willingness and ability of the participants to comply with the study protocol for the duration of the study.

Exclusion criteria

* For females: known pregnancy or breast feeding
* Participants who have received artemisinin or a derivative or an artemisinin-containing combination therapy (ACT) within the previous 7 days.
* History of allergy or known contraindication to artemisinins, lumefantrine or multivitamins
* Documented or claimed history of cardiac conduction problems
* Severe vomiting or diarrhoea
* Signs/symptoms of clinical malaria (febrile or history of fever in the previous 24 hours) confirmed by RDT.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1480 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of either clinical malaria with any Plasmodium species within 1-28, 29-56 or 57-84 days, or subclinical infection detected by PCR on days 28, 56 or 84. | 84 days

SECONDARY OUTCOMES:
28-day, 56-day, and 84-day PCR Plasmodium positivity rate for each species | 28, 56 and, 84 days
Proportion of participants with confirmed malaria reported between day 0 and day 28 for each species | 28 days
Incidence of confirmed clinical malaria cases as reported to government health facilities and village malaria workers.surveillance data. | 1 year
Prevalence of Kelch13 mutations and other genetic markers of antimalarial drug resistance of known functional significance. | 28 days
Incidence of adverse events and serious adverse events by study arms during the course of prophylaxis. | 28 days
a. Number of people living in each village b. Number of people working in each reported location c. Number of people who have travelled to different locations within the preceding 2 months d. Number of people who have a mobile phone for their own use | 28 days
Latitude and longitude of the study participant over time in decimal degrees as recorded every 10-30 minutes by a GPS logging device. | 28 days
Overall prevalence of Plasmodium at baseline, stratified by season and risk factors. | Day 0
Day 0, 28, 56 and 84 capillary blood levels of lumefantrine. | 84 days
Prevalence of serological diagnostic markers of other infectious diseases. | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Maude, M.D., Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (2):
- Cambodia (2):
  - Pursat Referral Hospital/Kravanh Health Center, Pursat
  - Stung Treng Referral Hospital/Siem Pang Health Center, Stung Treng

IPD SHARING:
Plan to Share IPD: Yes
De-identified, individual participant data from this study will be available to researchers whose proposed purpose of use is approved by the data access committee at Mahidol Oxford Tropical Medicine Research Unit. Inquiries or requests for the data may be sent to datasharing@tropmedres.ac.

REFERENCES:
- [Background] Guerra CA, Snow RW, Hay SI. A global assessment of closed forests, deforestation and malaria risk. Ann Trop Med Parasitol. 2006 Apr;100(3):189-204. doi: 10.1179/136485906X91512. PMID 16630376
- [Background] Thanh PV, Van Hong N, Van Van N, Van Malderen C, Obsomer V, Rosanas-Urgell A, Grietens KP, Xa NX, Bancone G, Chowwiwat N, Duong TT, D'Alessandro U, Speybroeck N, Erhart A. Epidemiology of forest malaria in Central Vietnam: the hidden parasite reservoir. Malar J. 2015 Feb 19;14:86. doi: 10.1186/s12936-015-0601-y. PMID 25880664
- [Background] Erhart A, Ngo DT, Phan VK, Ta TT, Van Overmeir C, Speybroeck N, Obsomer V, Le XH, Le KT, Coosemans M, D'alessandro U. Epidemiology of forest malaria in central Vietnam: a large scale cross-sectional survey. Malar J. 2005 Dec 8;4:58. doi: 10.1186/1475-2875-4-58. PMID 16336671
- [Background] Sanh NH, Van Dung N, Thanh NX, Trung TN, Van Co T, Cooper RD. Forest malaria in central Vietnam. Am J Trop Med Hyg. 2008 Nov;79(5):652-4. PMID 18981498
- [Background] Thang ND, Erhart A, Speybroeck N, Hung le X, Thuan le K, Hung CT, Ky PV, Coosemans M, D'Alessandro U. Malaria in central Vietnam: analysis of risk factors by multivariate analysis and classification tree models. Malar J. 2008 Jan 30;7:28. doi: 10.1186/1475-2875-7-28. PMID 18234102
- [Background] Erhart A, Thang ND, Hung NQ, Toi le V, Hung le X, Tuy TQ, Cong le D, Speybroeck N, Coosemans M, D'Alessandro U. Forest malaria in Vietnam: a challenge for control. Am J Trop Med Hyg. 2004 Feb;70(2):110-8. PMID 14993619
- [Background] Dysoley L, Kaneko A, Eto H, Mita T, Socheat D, Borkman A, Kobayakawa T. Changing patterns of forest malaria among the mobile adult male population in Chumkiri District, Cambodia. Acta Trop. 2008 Jun;106(3):207-12. doi: 10.1016/j.actatropica.2007.01.007. Epub 2008 Apr 7. PMID 18471797
- [Background] Moore SJ, Min X, Hill N, Jones C, Zaixing Z, Cameron MM. Border malaria in China: knowledge and use of personal protection by minority populations and implications for malaria control: a questionnaire-based survey. BMC Public Health. 2008 Oct 1;8:344. doi: 10.1186/1471-2458-8-344. PMID 18828901
- [Background] Gryseels C, Peeters Grietens K, Dierickx S, Xuan XN, Uk S, Bannister-Tyrrell M, Trienekens S, Ribera JM, Hausmann-Muela S, Gerrets R, D'Alessandro U, Sochantha T, Coosemans M, Erhart A. High Mobility and Low Use of Malaria Preventive Measures Among the Jarai Male Youth Along the Cambodia-Vietnam Border. Am J Trop Med Hyg. 2015 Oct;93(4):810-818. doi: 10.4269/ajtmh.15-0259. Epub 2015 Aug 17. PMID 26283747
- [Background] Grietens KP, Xuan XN, Ribera J, Duc TN, Bortel Wv, Ba NT, Van KP, Xuan HL, D'Alessandro U, Erhart A. Social determinants of long lasting insecticidal hammock use among the Ra-glai ethnic minority in Vietnam: implications for forest malaria control. PLoS One. 2012;7(1):e29991. doi: 10.1371/journal.pone.0029991. Epub 2012 Jan 12. PMID 22253852
- [Background] Lengeler C. Insecticide-treated bednets and curtains for preventing malaria. Cochrane Database Syst Rev. 2000;(2):CD000363. doi: 10.1002/14651858.CD000363. PMID 10796535
- [Background] Thang ND, Erhart A, Speybroeck N, Xa NX, Thanh NN, Ky PV, Hung le X, Thuan le K, Coosemans M, D'Alessandro U. Long-Lasting Insecticidal Hammocks for controlling forest malaria: a community-based trial in a rural area of central Vietnam. PLoS One. 2009 Oct 7;4(10):e7369. doi: 10.1371/journal.pone.0007369. PMID 19809502
- [Background] Son DH, Thuy-Nhien N, von Seidlein L, Le Phuc-Nhi T, Phu NT, Tuyen NTK, Tran NH, Van Dung N, Van Quan B, Day NPJ, Dondorp AM, White NJ, Thwaites GE, Hien TT. The prevalence, incidence and prevention of Plasmodium falciparum infections in forest rangers in Bu Gia Map National Park, Binh Phuoc province, Vietnam: a pilot study. Malar J. 2017 Nov 6;16(1):444. doi: 10.1186/s12936-017-2091-6. PMID 29110709
- [Background] York A. Seasonal malaria chemoprevention in the Sahel. Lancet Infect Dis. 2017 Jun;17(6):588. doi: 10.1016/S1473-3099(17)30255-4. No abstract available. PMID 28555586
- [Background] Snow RW. Seasonal Malaria Chemoprevention: An Evolving Research Paradigm. PLoS Med. 2016 Nov 22;13(11):e1002176. doi: 10.1371/journal.pmed.1002176. eCollection 2016 Nov. PMID 27875534
- [Background] Tripura R, Peto TJ, Chea N, Chan D, Mukaka M, Sirithiranont P, Dhorda M, Promnarate C, Imwong M, von Seidlein L, Duanguppama J, Patumrat K, Huy R, Grobusch MP, Day NPJ, White NJ, Dondorp AM. A Controlled Trial of Mass Drug Administration to Interrupt Transmission of Multidrug-Resistant Falciparum Malaria in Cambodian Villages. Clin Infect Dis. 2018 Aug 31;67(6):817-826. doi: 10.1093/cid/ciy196. PMID 29522113
- [Background] Imwong M, Hanchana S, Malleret B, Renia L, Day NP, Dondorp A, Nosten F, Snounou G, White NJ. High-throughput ultrasensitive molecular techniques for quantifying low-density malaria parasitemias. J Clin Microbiol. 2014 Sep;52(9):3303-9. doi: 10.1128/JCM.01057-14. Epub 2014 Jul 2. PMID 24989601
- [Background] Imwong M, Nguyen TN, Tripura R, Peto TJ, Lee SJ, Lwin KM, Suangkanarat P, Jeeyapant A, Vihokhern B, Wongsaen K, Van Hue D, Dong le T, Nguyen TU, Lubell Y, von Seidlein L, Dhorda M, Promnarate C, Snounou G, Malleret B, Renia L, Keereecharoen L, Singhasivanon P, Sirithiranont P, Chalk J, Nguon C, Hien TT, Day N, White NJ, Dondorp A, Nosten F. The epidemiology of subclinical malaria infections in South-East Asia: findings from cross-sectional surveys in Thailand-Myanmar border areas, Cambodia, and Vietnam. Malar J. 2015 Sep 30;14:381. doi: 10.1186/s12936-015-0906-x. PMID 26424000
- [Background] Saunders DL, Vanachayangkul P, Lon C; U.S. Army Military Malaria Research Program; National Center for Parasitology, Entomology, and Malaria Control (CNM); Royal Cambodian Armed Forces. Dihydroartemisinin-piperaquine failure in Cambodia. N Engl J Med. 2014 Jul 31;371(5):484-5. doi: 10.1056/NEJMc1403007. No abstract available. PMID 25075853
- [Background] West African Network for Clinical Trials of Antimalarial Drugs (WANECAM). Pyronaridine-artesunate or dihydroartemisinin-piperaquine versus current first-line therapies for repeated treatment of uncomplicated malaria: a randomised, multicentre, open-label, longitudinal, controlled, phase 3b/4 trial. Lancet. 2018 Apr 7;391(10128):1378-1390. doi: 10.1016/S0140-6736(18)30291-5. Epub 2018 Mar 29. PMID 29606364
- [Background] Bukirwa H, Unnikrishnan B, Kramer CV, Sinclair D, Nair S, Tharyan P. Artesunate plus pyronaridine for treating uncomplicated Plasmodium falciparum malaria. Cochrane Database Syst Rev. 2014 Mar 4;(3):CD006404. doi: 10.1002/14651858.CD006404.pub2. PMID 24596021
- [Background] Marks VA, Latham SR, Kishore SP. On Essentiality and the World Health Organization's Model List of Essential Medicines. Ann Glob Health. 2017 May-Aug;83(3-4):637-640. doi: 10.1016/j.aogh.2017.05.005. Epub 2017 Jun 22. PMID 29221540
- [Background] Agency, E.M., European Public Assessment Report for Pyramax. 2016.
- [Derived] Tripura R, von Seidlein L, Sovannaroth S, Peto TJ, Callery JJ, Sokha M, Ean M, Heng C, Conradis-Jansen F, Madmanee W, Peerawaranun P, Waithira N, Khonputsa P, Jongdeepaisal M, Pongsoipetch K, Chotthanawathit P, Soviet U, Pell C, Duanguppama J, Rekol H, Tarning J, Imwong M, Mukaka M, White NJ, Dondorp AM, Maude RJ. Antimalarial chemoprophylaxis for forest goers in southeast Asia: an open-label, individually randomised controlled trial. Lancet Infect Dis. 2023 Jan;23(1):81-90. doi: 10.1016/S1473-3099(22)00492-3. Epub 2022 Sep 26. PMID 36174595
- [Derived] Maude RJ, Tripura R, Ean M, Sokha M, Peto TJ, Callery JJ, Imwong M, Vongpromek R, Tarning J, Mukaka M, Waithira N, Soviet O, von Seidlein L, Sovannaroth S. Study protocol: an open-label individually randomised controlled trial to assess the efficacy of artemether-lumefantrine prophylaxis for malaria among forest goers in Cambodia. BMJ Open. 2021 Jul 7;11(7):e045900. doi: 10.1136/bmjopen-2020-045900. PMID 34233975

DOCUMENTS (2):
  • Study Protocol (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT04041973/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT04041973/SAP_001.pdf